CLINICAL TRIAL: NCT00446381
Title: Effect of Macugen (Pegaptanib) on Surgical Outcomes and Growth Factors Including Vascular Endothelial Growth Factor (VEGF) Levels in Patients With Proliferative Diabetic Retinopathy (PDR) and Clinically Significant Diabetic Macular Edema (CSDME)
Brief Title: Effect of Macugen(Pegaptanib)on Surgical Outcomes and VEGF Levels in Diabetic Patients With PDR (Diabetic Retinopathy or CSDME (Macular Edema)
Acronym: PEGAP001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Thomas G. Sheidow, MD, FRCSC, Ophthalmologist, Vitreoretinal Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R-06-821; Health Canada Control #108753
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Proliferative Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Proliferative Diabetic Retinopathy; Clinically Significant Diabetic Macular Edema; VEGF; Macugen (pegaptanib)
MeSH Terms: interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with Proliferative Diabetic Retinopathy
  Interventions: Drug: Macugen (pegaptanib)
- 2 (Experimental): Patients with Clinically Significant Macular Edema
  Interventions: Drug: Macugen (Pegaptanib)

INTERVENTIONS:
Drug: Macugen (pegaptanib) — Pegaptanib 0.3 mg by intravitreal injection once pre-operatively
  Arms: 1
Drug: Macugen (Pegaptanib) — Pegaptanib 0.3 mg by intravitreal injection once pre-operatively.
  Arms: 2

SUMMARY:
Patients with proliferative diabetic retinopathy or clinically significant diabetic macular edema requiring surgical intervention will receive a pre-operative injection of Macugen. An initial, pre-injection vitreous tap will be done in order to provide baseline VRGF 165 and cytokine levels. At the onset of the vitrectomy, a second vitreous sample will be taken to obtain intra-operative levels of Macugen, VEGF 165 and cytokines.

DETAILED DESCRIPTION:
Diabetes is one of the leading causes of blindness in North America. Diabetic retinopathy (PDR) is characterized by disruption of the normal microvascular circulation in the retina and results in the production of neovascularization and increased microvascular permeability. Similarly, clinically significant diabetic macular edema CSDME) results in loss of central visual acuity.

Many patients with these conditions, despite treatment, will go on to develop vitreous hemorrhage or tractional changes that require surgical intervention (such)as vitrectomy and/or vitrectomy with membrane peeling in the attempt to both restore vision and prevent further visual loss or re-establish the normal macular anatomy and improve patient visual acuity.

Although multiple etiologic factors are involved in the early changes seen in diabetic retinopathy and maculopathy, it has been shown that VEGF is the primary angiogenic growth factor implicated in the development of neovascularization in PRD and in increased vascular permeability, resulting in CSDME. VEGF levels have been found to correlate tightly with the extent of diabetic retinopathy and introduction of VEGF into normal primate eyes can induce diabetic retinopathy. Although several isoforms of VEGF exist, isoform 165 (VEGF 165) is the most pathogenic form of VEGF and therefore inhibition of VEGF 165 may play a significant role in modulating diabetic retinopathy and maculopathy.

Macugen is a VEGF antagonist (anti-VEGF pegylated aptamer) which binds to VEGF 165 with high specificity and affinity. In vitro pharmacology studies have shown that Macugen binds to the amino acid isoform VEGF 165 and inhibits it from binding to its cellular receptors. As a consequence, Macugen blocks signalling events and disrupts the cascade of proliferative and vascular permeability responses associated with the binding of VEGF 165 to endothelial cells. This effect has been clearly proven in Phase 3 trials for patients with age-related macular degeneration (AMD), resulting in inhibition of vascular development and decrease in vascular leakage.

Although diabetic retinopathy represents a different challenge than AMD, the underlying pathogenic factors are similar in the role and effects of VEGF. Regression of retinal neovascularization after Macugen therapy in diabetic individuals has been shown. Phase 2 studies have been completed and Phase 3 studies are currently underway in patients with diabetic macular edema to evaluate the efficacy of Macugen to restore vision in patients with CSDME. These studies are ongoing but exclude patients in whom vitrectomy has been performed or is planned in the near future due to tractional effects on the macula from epiretinal membranes or vitreomacular traction syndrome. No studies have been done to date in patients with PDR or CSDME to quantify the reduction of intravitreal VEGF 165 levels in these patients following intravitreal Macugen injection or to evaluate the effects of VEGF 165 blockade on the neovascular regression and surgical outcome in patients with extensive diabetic proliferative neovascularization.

The goal of this study is to quantify the reduction of intravitreal VEGF 165 levels in patients following intravitreal Macugen injection pre-operatively and determine the level of Macugen in the vitreous cavity after variable time intervals (2,4, 6 or 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Type 1 or 2 diabetes
* patients requiring surgical intervention for complications of proliferative diabetic retinopathy with vitreous hemorrhage or traction retinal detachment or clinically significant macular edema
* women postmenopausal for 12 months before the study, surgically sterile, or not pregnant and on effective contraception.

Exclusion Criteria:

* previous retinal vein occlusion.
* any intraocular surgery within the previous 12 months.
* myopia of > or = to 8 diopters.
* active ocular or periocular infection
* treatment with an investigational agent for any condition 60 days prior to enrollment.
* evidence of severe cardiac disease.
* clinically significant peripheral vascular disease (previous surgery, amputation, or symptoms of claudication)
* uncontrolled hypertension (treated systolic blood pressure > 155 mmHg or diastolic blood pressure > 95 mmHg)
* stroke within the preceding 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Levels of intravitreal Macugen post injection of intravitreal Macugen. | 2 to 8 weeks
Levels of intravitreal VEGF 165 pre and post injection of intravitreal Macugen. | 0 to 8 weeks
Levels of intravitreal VEGF, TGFbeta, ET-1, PDGF, IGF-1,angiopoietin, HIF 1 alpha, HIF 1 beta pre and post injection of intravitreal Macugen. | 0 to 8 weeks

SECONDARY OUTCOMES:
Effect on ease of surgery post injection of intravitreal Macugen. | 2 to 8 weeks
Effect on re-bleed rate post injection of intravitreal Macugen. | 0 to 8 weeks
Effect on concomitant diabetic macular edema post injection of intravitreal Macugen | 0 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Sheidow, MD, Principal Investigator — Ivey Eye Institute, St. Joseph's Health Care Centre
Locations (1):
- Ivey Eye Institute, St. Joseph's Health Care Centre, London, Ontario, Canada